CLINICAL TRIAL: NCT06600737
Title: Greater Manchester CARDIOvascular Pathology in Immune-Mediated Inflammatory Diseases
Acronym: GM CARDIO-IMID
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Prof. Maya H. Buch, Professor of Rheumatology and Director of Experimental Medicine at the Centre for Musculoskeletal Research, University of Manchester, University of Manchester
Other Study IDs: 320989
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cardiovascular Diseases; Rheumatologic Disease
MeSH Terms: conditions — Cardiovascular Diseases; Collagen Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — In total, 5 blood tubes (x1 plasma, x1 serum and x3 EDTA tube) will be collected, but if the maximum 75mls is needed additional blood tubes will be used. The blood samples may include peripheral blood mononuclear cells. Patients will have the opportunity to consent separately to a genetic (DNA) component. These samples will be collected during a participant's routine clinical appointment at the hospital by their clinical care or research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Disease Control (IMID and no CV disease): Control subjects will be asked to consent to a limited routine clinical, laboratory and imaging assessment and separate consent will be sought for imaging and biological sample collection. Consent for genetic (DNA) sample collection will be sought separately also.
  Where indicated, two groups of disease control patients will be recruited: (i) patients with an IMID and no CV disease and (ii) patients with CVD and no IMID diagnosis.
  The following assessments will be conducted (if indicated as part of a participants standard care):
  Clinician Questionnaires
  Clinical/medical, health and social care and social determinants
  Routine laboratory assessments
  Routine cardiovascular imaging and electrophysiology assessments
  Investigations to evaluate for cardiac conduction abnormalities and arrythmia may also be performed as part of routine care
  Routine peripheral vascular imaging assessment
  Patient reported outcome measures (PROMs) Questionnaires
- Disease Control (CV disease and no IMID): Control subjects will be asked to consent to a limited routine clinical, laboratory and imaging assessment and separate consent will be sought for imaging and biological sample collection. Consent for genetic (DNA) sample collection will be sought separately also.
  Where indicated, two groups of disease control patients will be recruited: (i) patients with an IMID and no CV disease and (ii) patients with CVD and no IMID diagnosis.
  The following assessments will be conducted (if indicated as part of a participants standard care):
  Clinician Questionnaires
  Clinical/medical, health and social care and social determinants
  Routine laboratory assessments
  Routine cardiovascular imaging and electrophysiology assessments
  Investigations to evaluate for cardiac conduction abnormalities and arrythmia may also be performed as part of routine care
  Routine peripheral vascular imaging assessment
  Patient reported outcome measures (PROMs) Questionnaires
- Healthy Control (no IMID history or CV disease): Control subjects will be asked to consent to a limited routine clinical, laboratory and imaging assessment and separate consent will be sought for imaging and biological sample collection. Consent for genetic (DNA) sample collection will be sought separately also.
  Healthy Control participants will have a limited number of assessments performed which may include:
  * Demographics, employment
  * Medical history, diagnoses, co-morbidities, symptoms, signs, lifestyle (smoking status (pack years) and alcohol intake (units/week), CVD risk scores
  * Detailed family history of autoimmune, vascular and rheumatic disease
  * Medications, vaccinations
  * Physical status (e.g. height and weight, blood pressure), IMID disease activity assessment as indicated
  * Data on hospital attendances and admissions, MACE, death registry information.
- Main Study (IMID 'at risk' CVD): Individuals who have a risk of developing CVD (based on traditional risk factors and/or IMID-specific factors) but no history of major adverse cardiovascular events (MACE).
  The main study represents standard clinical care and includes the routine clinical, laboratory and imaging assessments. Patients may be recruited at any point along their CVD continuum (eg when considered at risk, at time of or after a diagnosis of a CVD).
  The following assessments will be conducted (if indicated as part of a participants standard care):
  Clinician Questionnaires
  Clinical/medical, health and social care and social determinants
  Routine laboratory assessments
  Routine cardiovascular imaging and electrophysiology assessments
  Investigations to evaluate for cardiac conduction abnormalities and arrythmia may also be performed as part of routine care
  Routine peripheral vascular imaging assessment
  Patient reported outcome measures (PROMs) Questionnaires
- Main Study (Incident (new) IMID-CVD): Patients with IMID that present with a MACE.
  The main study represents standard clinical care and includes the routine clinical, laboratory and imaging assessments. Patients may be recruited at any point along their CVD continuum (eg when considered at risk, at time of or after a diagnosis of a CVD).
  The following assessments will be conducted (if indicated as part of a participants standard care):
  Clinician Questionnaires
  Clinical/medical, health and social care and social determinants
  Routine laboratory assessments
  Routine cardiovascular imaging and electrophysiology assessments
  Investigations to evaluate for cardiac conduction abnormalities and arrythmia may also be performed as part of routine care
  Routine peripheral vascular imaging assessment
  Patient reported outcome measures (PROMs) Questionnaires
- Main Study (Established IMID-CVD): Patients with IMID and a history of previous MACE.
  The main study represents standard clinical care and includes the routine clinical, laboratory and imaging assessments. Patients may be recruited at any point along their CVD continuum (eg when considered at risk, at time of or after a diagnosis of a CVD).
  The following assessments will be conducted (if indicated as part of a participants standard care):
  Clinician Questionnaires
  Clinical/medical, health and social care and social determinants
  Routine laboratory assessments
  Routine cardiovascular imaging and electrophysiology assessments
  Investigations to evaluate for cardiac conduction abnormalities and arrythmia may also be performed as part of routine care
  Routine peripheral vascular imaging assessment
  Patient reported outcome measures (PROMs) Questionnaires
- Imaging Sub-Study: In addition to the main study, patients will be offered the opportunity to consent to participate in the imaging Sub-Study.
  Patients consenting to the Imaging Sub-Study must also have consented to participate in the Main Study. Assessments conducted as part of the Main Study are outlined in the relevant 'Main Study' Group/Cohort descriptions.
  Individuals participating in the Imaging Sub-Study may be asked to undergo additional imaging tests above standard of care (undertaken separately to the main study assessments/visits) using dedicated research protocols.
  The following assessments may be conducted:
  Echocardiography
  Cardiovascular Magnetic Resonance Imaging (CMR)
  Peripheral vascular imaging techniques:
  Laser Doppler Imaging (LDI) and laser speckle contrast imaging (LSCI)
  Nailfold capillaroscopy
  Multispectral imaging
  Non-vascular skin imaging techniques:
  High frequency ultrasound
- Biological Sub-Study: In addition to the Main Study, patients will be offered the opportunity to consent to participate in the Biological Sub-Study.
  Patients consenting to the Biological Sub-Study must also have consented to participate in the Main Study. Assessments conducted as part of the Main Study are outlined in the relevant 'Main Study' Group/Cohort descriptions.
  Biological samples as part of the Sub-Study are in addition to standard of care blood samples.
  A maximum of 75mls of blood may be taken to enable the range of experimental studies. The samples may be taken at initial time of recruitment (baseline) and/or may be repeated at certain time points depending on the diagnosis and if a change in the clinical status (excluding genotyping).
  The blood may be drawn into a combination of EDTA, lithium heparin, red clotted, citrate and PAXGENE/TEMPUS tubes, according to planned experiments at each time point.

SUMMARY:
The researchers would like to know more about cardiovascular abnormalities in patients with immune-mediated inflammatory diseases (IMID) and with the aim to provide new biomarkers (clinical, blood, imaging) for early diagnosis, prognosis and prediction of CVD in patients with IMID. This is important as there are still many things that are not known about this and finding out more could improve how patients are treated in future.

Participants with IMID diagnoses will be recruited from rheumatology/cardiology departments as in-patients or outpatients.

Once consented, researchers will collect past, present and future clinical information about them, including routine cardiovascular imaging and blood tests. Participants will also be asked to complete questionnaires at predetermined intervals. The participants could also be approached to take part in the following sub-studies; Biological sub-study, in which blood and urine would be collected; And the Imaging-sub study, in which one or more of Echocardiography, Cardiovascular Magnetic Resonance Imaging (CMR) and Laser Doppler Imaging (LDI) will be performed. Participants with CVD without IMID and healthy volunteers will also be recruited as comparison groups.

The research is to be funded by the NIHR Manchester BRC ('Integrated Cardiovascular' and 'Rheumatic & Musculoskeletal Diseases' themes). Other funding eg Manchester Academic Health Sciences and a recently awarded Medical Research Council Partnership grant will also support this programme. The study will recruit in specialist NHS centres; Recruitment will start in Manchester University Hospitals NHS Foundation Trust.

DETAILED DESCRIPTION:
Immune-mediated-inflammatory-diseases (IMID) are a range of illnesses affecting over 1 million people in the UK.

Targeted treatments have changed outcomes of common IMIDs, but mortality is still high, largely due to premature cardiovascular disease (CVD). IMID includes the common rheumatoid arthritis (RA), systemic lupus erythematosus (SLE) and related conditions, and rare diseases such as systemic sclerosis (SSc), idiopathic inflammatory myopathies (IIM) and vasculitides. Increased risk of CVD and death in IMID contributes to inflammation and cardio metabolic disorders which includes accelerated atherosclerosis, microvascular dysfunction and myocardial and pericardial disease. The research has shown people with RA have a 50% higher risk for CVD than the general population and up to 35% of deaths in patients with SSc are due to cardiac causes.

The biological mechanisms underlying CVD in IMIDs remain largely unknown. Two comparable IMID patients may have significant differences in the presence of CVD and the reasons for this are poorly understood. Despite the significant morbidity and mortality associated with CVD in IMID patients, identification of at-risk patients early in the disease to start treatments and improve prognosis remains challenging. Difficulties also persist in tailoring treatments for people with IMID and existing CVD and there is an evidence gap in treating certain kind of cardiovascular involvement for example, myocarditis. This proposed study will address the missing gaps of the current knowledge. The longitudinal collection and evaluation of routine clinical information and imaging data at different stages of disease will allow the researchers to develop a prognostic model to identify risk factors for CVD in IMID and identify at-risk IMID patients. In addition, the biological and imaging sub-studies will allow the researchers to gain comprehensive insights into the mechanisms underlying CVD in IMID patients, including molecular pathways, genetics and imaging biomarkers. This programme of work will generate important pilot data that will inform subsequent definitive and fully powered studies.

Any potentially eligible patients seen at the relevant rheumatology/cardiology departments as part of in-patient, outpatient and/or multi-disciplinary team meetings and identified as per usual clinical practice may be eligible for inclusion in this observational programme; these patients will be classified as IMID patients at-risk of CVD (IMID-'at risk' CVD), IMID patients with documented new major adverse cardiovascular event (MACE) (Incident IMID-CVD) and IMID patients with previous MACE (Established IMID-CVD). Three groups of control patients will also be recruited; IMID patients with no risk of CVD, patients with CVD but no IMID diagnosis and healthy volunteers.

The doctor will explain to the patient about the study and, if they are interested provide them with the information leaflet.

The participant will have the opportunity to ask the research staff questions after they have seen the paperwork.

Patients may consent same day and/or be given the opportunity to discuss the trial with their family before they are asked whether they would be willing to take part in the trial. If English is not the patient's first language every effort will be made to provide a Trust interpreter according to normal Trust procedures. This is an observational longitudinal study where past, present and future routine clinical data and tests (such as hospital presentations, blood tests, imaging) and/or additional sub-study specific research data will be collected and entered into a database. Following consent, data will be obtained as per usual clinical visits and assessments.

Patients are seen as per standard clinical practice determined by the index IMID and in this setting, also dependent on co-existing CV comorbidity. This would usually be every 6 months at time of IMID/CVD diagnosis and then 12 monthly thereafter. Following consent, data from before this time point may be obtained through the available health records.

Participants will also be asked to complete questionnaires determined by their IMID diagnosis and/or CVD profile at follow up appointments. These will be returned to the University of Manchester along with a registration form that will include confirmation of a participant's contact information. Patients will be given the opportunity to consent to the biological and/or imaging sub-studies. Unlike the main study, participants will be asked to undergo biological tests (blood tests or urine sample if applicable) or imaging tests (echocardiography, cardiac magnetic resonance imaging, peripheral imaging) in addition to routine standard care.

Where possible, these additional tests will be combined with routine clinical care to minimise inconvenience to the participant, for example collecting additional blood tests at same time of routine clinical blood test. The additional imaging studies would need to be done on a separate visit to the routine clinical follow up.

All procedures will be carried out by their local NHS clinical or research team at the Unit they are normally seen in MFT (MRI/Wythenshawe site) based on usual site of care, and will be carried out by trained staff. This is designed to fit around standard care as much as possible and provide as little inconvenience as possible to potential participants.

All control subjects will be treated in the same way patient participants are; The face-to-face consent process will be the same. The research team will explain what is required of them, what procedures they would be undertaking, and the detail of these and where they would occur. Patient-reported outcomes relevant to the IMID and/or CVD profile may be taken at each visit, if the participant consents to this. These may include RAQoL, HAQ, EQ-5D, ScleroID and clinician assessed New York Heart Association (NYHA) classification (based on the patient history). The research staff at the recruiting centre will access participant's medical records, where consent is provided for them to do so. They will enter appropriate research data into an electronic case report form (eCRF) on the hospital site. In the eCRF, participants will be identified by study number only. No personal identifiable information (PII) will be included in the eCRF.

ELIGIBILITY:
Main Study

Inclusion Criteria:

* Males and females
* Subjects aged over 18 years
* Capable of providing informed consent and signing a consent form
* Have a clear diagnosis of an IMID with history consistent with one of the following categories:
* IMID-'at risk' CVD: individuals who have a risk of developing CVD (based on traditional risk factors and/or IMID-specific factors) but no history of major adverse cardiovascular events (MACE).
* Incident (new) IMID-CVD: Patients with IMID that present with a MACE.
* Established IMID-CVD: Patients with IMID and a history of previous MACE

Exclusion Criteria:

* Age less than 18 years
* Lack of capacity to give informed consent

Imaging Sub-Study

Inclusion Criteria:

- As-listed for Main Study

Exclusion Criteria:

* As-listed for Main Study and;
* For the research cardiac MRI imaging component, the following exclusions will apply: pacemakers, surgical clips within the head, certain inner ear implants, neuro-electrical stimulators or metal fragments within the eye or head, pregnancy or breast-feeding. For administration of gadolinium-based contrast agent, GFR < 30 ml/min/1.73 m2 is a contraindication.

Biological Sub-Study

Inclusion Criteria:

- As-listed for Main Study

Exclusion Criteria:

- As-listed for Main Study

Controls

Inclusion Criteria:

* Subject ≥ 18 years of age
* Is capable of understanding and signing an informed consent form
* No known diagnosis of an IMID (CVD-no IMID disease control and healthy control groups)
* No known diagnosis of CVD (IMID-no risk CVD disease control and healthy control groups)

Exclusion Criteria:

* As-listed for Main Study and;
* For the research cardiac MRI imaging component, the following exclusions will apply: pacemakers, surgical clips within the head, certain inner ear implants, neuro-electrical stimulators or metal fragments within the eye or head, pregnancy or breast-feeding. For administration of gadolinium-based contrast agent, GFR < 30 ml/min/1.73 m2 is a contraindication.

For Healthy controls:

The researchers will aim to identify healthy controls using the 'bring a friend' strategy where the patient is asked to bring a friend/relative, thus minimising demographic bias. This will establish a healthy control pool. For specific analyses, controls will be age and sex matched and where possible, BMI-matched to the specific study population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from NHS secondary care in the United Kingdom. Potential participants may be identified from clinics, wards, diagnostic pathways and departments, electronic and paper-based health records, databases and waiting lists in secondary care. All individuals will be considered for inclusion in this study regardless of age, disability, gender reassignment, marriage and civil partnership, pregnancy and maternity, race, religion and belief, sex, and sexual orientation, except where the study inclusion and exclusion criteria explicitly state otherwise.
Sampling Method: Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2032-09-01 (Estimated); Study Completion 2032-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with major adverse cardiovascular events (MACE) | 10 Years
  Major Adverse Cardiovascular Events (MACE) is a grouped term typically defined as acute myocardial infarction, stroke or cardiovascular death. Primary myocardial events such as myocarditis (especially relevant to IMIDs such as SSc, IIM, SLE) will also form part of the primary MACE definition.
  The total number of participants presenting with or developing a MACE will be measured.
  Unit: number of participants

SECONDARY OUTCOMES:
Number of participants with heart failure hospitalisations | 10 Years
  Extended MACE endpoints that may comprise all ischaemic CV events/significant clinical outcomes will also be captured: Heart failure hospitalisation, unstable angina, need for revascularisation, all-cause mortality.
  The total number of participants hospitalised with heart failure will be measured.
  Unit: number of participants
Number of participants with unstable angina | 10 Years
  Extended MACE endpoints that may comprise all ischaemic CV events/significant clinical outcomes will also be captured: Heart failure hospitalisation, unstable angina, need for revascularisation, all-cause mortality.
  The total number of participants with unstable angina will be measured.
  Unit: number of participants
Number of participants needing revascularisation | 10 Years
  Extended MACE endpoints that may comprise all ischaemic CV events/significant clinical outcomes will also be captured: Heart failure hospitalisation, unstable angina, need for revascularisation, all-cause mortality.
  The total number of participants needing revascularisation will be measured.
  Unit: number of participants
Number of participants with abnormal high-sensitivity cardiac troponin I/T levels | 10 Years
  The total number of participants with abnormal high-sensitivity troponin I/T levels (assessed by blood draw) will be measured.
  Unit: number of participants
Number of participants with abnormal ECHO and or CMR imaging measures | 10 Years
  ECHO and or CMR imaging measures include atrial and ventricular volumetrics, systolic and diastolic function, regional wall motion abnormalities, myocardial inflammation (CMR only), presence and extent of replacement fibrosis (CMR only), aortic distensibility (CMR only).
  The total number of participants with abnormal ECHO and/or CMR imaging measures will be measured.
  Unit: number of participants
Number of participants with abnormal N-terminal pro B-type natriuretic peptide (NT-pro BNP) levels | 10 Years
  The total number of participants with abnormal NT-pro BNP levels (assessed by blood draw) will be measured.
  Unit: number of participants
Number of participants with abnormal Creatine Kinase (CK) levels | 10 Years
  The total number of participants with abnormal Creatine Kinase levels (assessed by blood draw) will be measured.
  Unit: number of participants

CONTACTS AND LOCATIONS:
Overall Officials: Maya H Buch, MD, Principal Investigator — University of Manchester
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom